CLINICAL TRIAL: NCT00483743
Title: Multi-Center, Randomized, Double-Blind, Placebo and Active-Controlled, 6-week Study to Evaluate the Safety, Tolerability and Pharmacodynamic Activity of Inhaled TPI 1020 in COPD Patients.
Brief Title: Safety, Tolerability and PD Activity of Inhaled TPI 1020 Versus Inhaled Budesonide in COPD Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Syntara (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TPI 1020-203
Record Dates: First submitted 2007-05-23; First posted 2007-06-07 (Estimated); Last update posted 2012-12-03 (Estimated); Status verified 2012-11

CONDITIONS: Copd Bronchitis
MeSH Terms: interventions — NCX 1020; Budesonide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- TPI 1020 (Experimental): TPI 1020 500 mcg BID x 42 days
  Interventions: Drug: TPI 1020
- Budosenide cortico (Active Comparator): Budesonide 800 mcg BID x 42 days
  Interventions: Drug: Budesonide
- Placebo (Placebo Comparator): Placebo inhaler
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TPI 1020 — 250 mcg/caps 2 caps BID x 42 days
  Arms: TPI 1020
Drug: Budesonide — 400mcg mcg capsules- 2 capsules BID
  Arms: Budosenide cortico
Drug: Placebo — 2 caps BID x42 days
  Arms: Placebo

SUMMARY:
This study will assess and compare the safety and tolerability of inhaled TPI 1020 (repeated nominal doses; 500 μg BID x 6 weeks) versus inhaled budesonide (repeated doses; 800 μg BID x 6 weeks) and a matching placebo. Pharmacodynamic (PD) activity on FEV1, sputum and blood cells and cytokines will also be studied.

DETAILED DESCRIPTION:
A multi-centre, randomized, placebo and active-controlled, 6-week study of inhaled TPI 1020, inhaled budesonide or matching placebo (random allocation of eligible patients to the three treatments at a ratio of 3:3:1), to evaluate the safety, tolerability and pharmacodynamic activity of TPI 1020 in 42 evaluable COPD subjects.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients, male or female, smoker or ex-smoker (who quit at least a year ago) with a smoking history equal or greater than 10 pack years.
* Age between 40 and 80 years old with a diagnosis (for at least 12 months) of mild to moderate COPD

Exclusion Criteria:

* COPD exacerbations indicated by a treatment with oral or systemic glucocorticosteroids and/or hospitalization and/or clinically relevant respiratory infection requiring antibiotics within 3 month of the start of the study.
* Failure to produce a sufficient sputum sample during the screening sputum induction procedure, required for TCC and differential cell count determination.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2007-11; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
To determine the airway specific, and general safety and the tolerability of inhaled TPI 1020 administered via Aerolizer™ in COPD patients. • To assess the effects of TPI 1020 versus those of budesonide on sputum neutrophil counts on Days 0 and 42. | 42 days

SECONDARY OUTCOMES:
Sputum neutrophil counts on Days 0 and 21. • Trough FEV1, SVC and IC on Days 0, 21 and on Day 42. • eNO levels on Days 0, 21 and on Day 42. | 42 days

CONTACTS AND LOCATIONS:
Overall Officials: Francois Maltais, MD, Principal Investigator — Centre de Cardiologie et de Pneumologie de l'Université Laval; Rene Pageau, M.Sc Pharm, Study Director — Syntara
Locations (13):
- Canada (13):
  - University of alberta Hsopital, Edmonton, Alberta
  - Vancouver Hospital Lung Center, Vancouver, British Columbia
  - Firestone Institute for Respiratory Health, Hamilton, Ontario
  - Clinique Medical Les Saules, Les Saules, Quebec
  - Omnispec Clinical Research Inc., Mirabel, Quebec
  - Hopital Thoracique Montreal-CSUM, Montreal, Quebec
  - Hopital Sacre Coeur de Montreal, Montreal, Quebec
  - Kells Medical Research Group, Pointe-Claire, Quebec
  - Complexe Medicale Langelier, Saint-Léonard, Quebec
  - Diex Research Inc., Sherbrooke, Quebec
  - CHUS -Hopital FLEURIMONT, Sherbrooke, Quebec
  - Centre de Cardiologie et de Pneumologie de l'Université Laval, Ste-Foy, Quebec
  - Royal University Hospital, Saskatoon, Saskatchewan